CLINICAL TRIAL: NCT02909634
Title: Combining Ostom-I With Abstats Sensors to Improve Prediction of Ostomy Output
Status: Withdrawn | Type: Observational
Why Stopped: No devices currently available for study.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: 11 Heath and Technologies Limited (Industry)
Responsible Party: Principal Investigator, Christopher Almario, Health Services Research Scientist, Cedars-Sinai Medical Center
Other Study IDs: Pro00046068
Record Dates: First submitted 2016-09-14; First posted 2016-09-21 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Ostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, the number of patients having either permanent or temporary stomas placed is increasing each year. Yet, patients with ostomy pouches often struggle with predicting when stool output will occur and how to plan around dynamic changes in intestinal activity. Ostom-I provides a real-time assessment of the volume in the ostomy bag, it does not predict when and how fast such output will occur. In this pilot study the investigators aim to gather normative AbStats and Ostom-I data in participants with an ostomy to improve prediction of stool output.

Aim 1: To gather normative AbStats and Ostom-I data in subjects with an ostomy to improve prediction of stool output.

Aim 2: Correlate the data from both wearable biosensors and test the predictive validity of AbStats in determining ostomy bag filling as measured by Ostom-I.

DETAILED DESCRIPTION:
The Ostom-I device is a wireless, wearable biosensor that is approved by the U.S. Food and Drug Administration (FDA). The device is discrete, lightweight, and can be applied to an ostomy pouch in order to monitor the filling of the bag. It uses Bluetooth technology to send a signal to the participants smartphone and alerts the user when the ostomy bag is filling up so they can decide if and when to empty them.The second wearable biosensor is called "AbStats" and it provides an objective, real-time marker of intestinal motility, and is also FDA approved. It allows for continuous and automated analysis of intestinal vibrations.The study team will recruit consecutive inpatients undergoing colorectal surgery with ostomy placement. The surgeon will apply AbStats and Ostom-I upon completion of the operation. Device recordings will continue until discharge, or until the participant opts to remove the sensors as requested. Members of the research team who are blinded to sensor results will monitor and record clinical information including age, gender, race, and body mass index (BMI). The study team will record type of surgery performed, surgical approach, and any documented operative complications. The study team will prospectively monitor daily clinical assessments, including symptoms (nausea, vomiting, and abdominal pain), flatus, bowel movements, diet, ambulation, medication use, and length of hospitalization. All patients will receive a standardized feeding protocol as part of usual care. For Cedars-Sinai, the standard protocol initiates clear liquids on postoperative day (POD) zero, and rapid progression to a regular diet by the morning of POD#1 in patients without early clinical evidence of post-operative ileus (POI). Patients intolerant of the feeding protocol, including nausea or vomiting precluding advancement, or those that develop significant abdominal distension, will discontinue the feeding protocol. The surgical teams that make the decisions regarding diet changes will be blinded to device data.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing abdominal surgery
* Able to provide informed consent

Exclusion Criteria:

* Unable to provide consent
* Cognitive inability to follow directions to maintain sensors in place
* Unable to place abdominal sensors on patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients undergoing colorectal surgery with ostomy placement
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Average intestinal rates needed to fill 1/4 and 1/2 of ostomy pouch | Preceding 5 hours
  Defined as area under the curve for a plot of intestinal rate vs. time
Max intestinal rate following 1/4 and 1/2 filling of the ostomy pouch | Preceding 5 hours
  Defined as maximum intestinal rate achieved in preceding 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christopher V Almario, MD, MSHPM, Principal Investigator — Cedars-Sinai Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spiegel BM, Kaneshiro M, Russell MM, Lin A, Patel A, Tashjian VC, Zegarski V, Singh D, Cohen SE, Reid MW, Whitman CB, Talley J, Martinez BM, Kaiser W. Validation of an acoustic gastrointestinal surveillance biosensor for postoperative ileus. J Gastrointest Surg. 2014 Oct;18(10):1795-803. doi: 10.1007/s11605-014-2597-y. Epub 2014 Aug 5. PMID 25091837
- [Background] Kaneshiro M, Kaiser W, Pourmorady J, Fleshner P, Russell M, Zaghiyan K, Lin A, Martinez B, Patel A, Nguyen A, Singh D, Zegarski V, Reid M, Dailey F, Xu J, Robbins K, Spiegel B. Postoperative Gastrointestinal Telemetry with an Acoustic Biosensor Predicts Ileus vs. Uneventful GI Recovery. J Gastrointest Surg. 2016 Jan;20(1):132-9; discussion 139. doi: 10.1007/s11605-015-2956-3. Epub 2015 Sep 25. PMID 26408329